CLINICAL TRIAL: NCT01454531
Title: An Open Trial to Assess the Tolerability of AVANZ Phleum Pratense Immunotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-G-01
Record Dates: First submitted 2011-10-13; First posted 2011-10-19 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Rhinoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVANZ Phleum pratense (Experimental): AVANZ Phleum pratense up-dosing phase (300, 600, 3000, 6000 and 15,000 SQ+) + one 15,000 SQ+ maintenance injection
  Interventions: Drug: AVANZ Phleum pratense

INTERVENTIONS:
Drug: AVANZ Phleum pratense — AVANZ Phleum pratense up-dosing phase (300, 600, 3000, 6000 and 15,000 SQ+) + one 15,000 SQ+ maintenance injection

SUMMARY:
The purpose of this study is to assess the tolerability of AVANZ.

DETAILED DESCRIPTION:
To assess the tolerability of the up-dosing phase of AVANZ Phleum pratense. The frequency of patients with adverse reactions will be the study primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* History of grass pollen rhinoconjunctivitis
* Positive SPT to Phleum pratense
* Positive specific IgE against Phleum pratense

Exclusion Criteria:

* Uncontrolled severe asthma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JOAQUIN SASTRE, MD, PhD, Principal Investigator — FUNDACIÓN JIMÉNEZ DIAZ
Locations (20):
- Spain (20):
  - Hospital de Basurto, Bilbao, Bilbao
  - Fundación Jiménez Diaz, Madrid, Madrid
  - Hospital Infanta Elena, Madrid, Madrid
  - Hospital Universitari Politecnic La Fe, Valencia, Valencia
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital Universitario Infanta Cristina, Badajoz
  - Complejo Hospitalario de Burgos, Burgos
  - Hospital Nuestra Señora de La Montaña, Cáceres
  - H. Campo Arañuelo, Cáceres
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Univesitario Fundación Hospital de Alcorcón, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Rio Carrion, Palencia
  - Hospital Santa Bárbara, Puertollano
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Univeritario Marques de Valdeilla, Santander
  - Hospital Santiago Apostol, Vitoria-Gasteiz
  - Hospital Virgen de La Concha, Zamora

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 199 subjects were recruited and 3 resulted screening failures so 196 subjects started the trial. Four subjects discontinued before treatment so 192 subjects were treated. The reason for discontinuation for these 4 subjects was withdrawal of consent ("Withdrawal by subject", included in Reasons Not Completed)
Groups:
- AVANZ Phleum Pratense: AVANZ Phleum pratense
  AVANZ Phleum pratense: Up-dosing phase of AVANZ Phleum pratense
Period: Overall Study
Arm/Group | AVANZ Phleum Pratense
Started | 196
Subjects Treated | 192
Completed | 173
Not Completed | 23
Not completed — Adverse Event | 14
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Delay in IMP administration | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Subjects treated
Arm/Group | AVANZ Phleum Pratense
Number analyzed (Participants) | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 94
Region of Enrollment [Number; unit: participants]
  Spain | 192

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Subjects With Adverse Drug Reactions
Description: Frequency of patients with adverse reactions, local or systemic
Time Frame: 6 weeks
Population: Subjects treated
Measure: Number; unit: participants
Arm/Group | AVANZ Phleum Pratense
Number analyzed (Participants) | 192
participants | 133

2. Secondary Outcome: Frequency of Subjects With Systemic Reactions
Description: Frequency of patients with systemic reactions, based on EAACI classification: Grade I (mild systemic reaction) to IV (anaphylactic shock)
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | AVANZ Phleum Pratense
Number analyzed (Participants) | 192
participants | 66

3. Secondary Outcome: Frequency of Subjects With Local Adverse Reaction
Description: Frequency of patients with local adverse reactions
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | AVANZ Phleum Pratense
Number analyzed (Participants) | 192
participants | 109

4. Secondary Outcome: Change in Phleum Pratense Specific IgE-blocking Factor
Description: IgE-blocking factor measures the amount of IgE bound to the allergen in the presence of allergen-competing factors present in the serum of a subject treated with allergen immunotherapy. The test is based in a double IgE measurement, an ordinary assay and an assay in the presence of competing components and takes the form of:
  IgE blocking factor = 1 - (Competitive IgE/Ordinary IgE). Theoretical limits are from 0 (no IgE blocked) to 1 (all IgE blocked) and, being a ratio, is a dimensionless measure
Time Frame: baseline (visit 1) and at 6 weeks (visit 6)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | AVANZ Phleum Pratense
Number analyzed (Participants) | 167
arbitrary units
  Visit 1 | -0.13 (0.2)
  Visit 6 | 0.12 (0.3)
Statistical Analysis 1: Comparison: AVANZ Phleum Pratense; The null hypothesis is no changes in IgE-blocking factor values from visit 1 (baseline) to visit 6 (end of treatment) versus the alternative hypothesis of change in IgE-blocking factor values; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Paired values

5. Secondary Outcome: Change in Phleum Pratense Specific IgG4
Time Frame: baseline (visit 1) and at 6 weeks (visit 6)
Population: Number of subject with valid data in visit 1 and visit 6
Measure: Mean (Standard Deviation); unit: mgA/l
Arm/Group | AVANZ Phleum Pratense
Number analyzed (Participants) | 171
mgA/l
  Visit 1 | 0.44 (0.6)
  Visit 6 | 2.26 (2.5)
Statistical Analysis 1: Comparison: AVANZ Phleum Pratense; The null hypothesis is no changes in Phleum specific IgG4 values from visit 1 (baseline) to visit 6 (end of treatment) versus the alternative hypothesis of change in Phleum specific IgG4 values; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Paired samples

6. Secondary Outcome: Change in Immediate Cutaneous Response to Phleum Pratense
Description: Wheal size provoked after prick test with 4, 20 and 100 µg/ml Phl p 5 allergen extracts analysed by Parallel Line Assay. Cutaneous Tolerance Index (CTI) is the factor it is necessary to multiply the extract concentration by after SCIT (V6) to obtain the same response in terms of wheal area as at baseline (V1). CTI, being an index, is a dimensionless measure. A CTI of 1 indicates no change in skin sensitivity while if higher than 1 a decrease in skin sensitivity (it would be needed a more concentrated allergen extract at V6 to elicit the same skin response as at V1
Time Frame: baseline (visit 1) and at 6 weeks (visit 6)
Population: Participants in which results of the Parallel Line Assay are valid
Measure: Mean (95% Confidence Interval); unit: CTI, Cutaneous Tolerance Index
Arm/Group | AVANZ Phleum Pratense
Number analyzed (Participants) | 129
CTI, Cutaneous Tolerance Index | 1.79 [1.49 to 2.16]
Statistical Analysis 1: Comparison: AVANZ Phleum Pratense; Parallel Line Assay is based on the construction of two dose-response regression lines obtained plotting the allergen concentration used to prick test the subjects against the wheal size obtained. ANOVA allows to check for regression, linearity and parallelism. A common slope and y-intercepts are calculated. The CTI is the exponentiation of the difference between y-intercepts divided by the common slope. (Finney D.J., Statistical Method in Biological Assay, 1978); Test type: Superiority or Other; p < 0.01, Parallel Line Assay

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | AVANZ Phleum Pratense
Serious Adverse Events (participants affected / at risk) | 3/192
Other Adverse Events (participants affected / at risk) | 109/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVANZ Phleum Pratense (N=192)
Generalised urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVANZ Phleum Pratense (N=192)
Hypersensitivity (Immune system disorders) | 10 (14)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 15 (19)
Urticaria (Skin and subcutaneous tissue disorders) | 17 (17)
Local reactions (General disorders) | 109 (262) — Includes injection site pain, erythema, pruritus and/or swelling of any intensity or size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All presentations/publications must be approved by ALK prior to public presentation/submission. Investigators agree not to present data gathered from one trial centre or a small group of trial centres before the full publication unless formally agreed by all other investigators and ALK. ALK has the right to review and comment any manuscript within 30 days of receipt, but cannot prevent publications of findings.